CLINICAL TRIAL: NCT03020693
Title: Effectiveness of Invasive Electrostimulation Combined With an Exercise Program in Plantar. A Clinical Trial
Brief Title: Effectiveness of Invasive Electrostimulation Combined With an Exercise Program in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-2015-12
Record Dates: First submitted 2016-12-28; First posted 2017-01-13 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-02

CONDITIONS: Fasciitis, Plantar
Keywords: electrostimulation; exercise program
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Exercise; Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive electrostimulation combined with exercises. (Experimental): Dry needling + TENS ( 4 Hz 200 microseconds during 30 minutes to therapeutic intensity) combined with exercises program.
  Interventions: Procedure: Invasive electrostimulation combined with exercises
- Placebo electrostimulation and exercises. (Active Comparator): Sham dry needling + TENS ( 4 Hz 200 microseconds during 30 minutes to non-therapeutic intensity) with surface electrodes combined with exercises program.
  Interventions: Procedure: Placebo electrostimulation and exercises

INTERVENTIONS:
Procedure: Invasive electrostimulation combined with exercises — Procedure for producing analgesia by introducing the TENS current through a needle combined with a exercises program.
  Other Names: dry needling with TENS
  Arms: Invasive electrostimulation combined with exercises.
Procedure: Placebo electrostimulation and exercises — First: Sham dry needling. After: electrostimulation using surfaces electrodes. Finally a exercises program.
  Other Names: Non-invasive electrostimulation combined with exercises
  Arms: Placebo electrostimulation and exercises.

SUMMARY:
This study evaluates the effectiveness of an electrostimulation treatment with TENS using a needle and a surface electrode combined with an exercise program to fasciitis plantar. Half participants will receive invasive electrostimulation (TENS using a needle) and exercises while the other half will receive electrostimulation placebo and exercises.

DETAILED DESCRIPTION:
There are a lot of treatments to fasciitis plantar. Exercises are the treatments more recommended to fasciitis plantar but not all patients improve only with exercises. Dry needling is recommended to relieve the pain in the heel. TENS is used to decrease the pain in the fasciitis plantar. Investigators will apply to half participants a treatment that combines TENS + Dry needling (invasive electrostimulation ) with exercises while the other half receive electrostimulation placebo (TENS using surface electrodes with non-therapeutic intensity) + exercises.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of plantar fasciitis
* Age equal or superior to 18 years old.
* VAS minimum of 2 points int the first steps after a prolonged decreasing period.
* Having an evolution of a month or more of pain.
* Not having received acupuncture or dry needling as treatment.

Exclusion Criteria:

* Peripheral Neuropathies.
* Tarsus tunnel syndrome.
* Rheumatic diseases.
* Contraindication to dry needling: nickel allergy, fear of needles, sky with erosions.
* Clotting disorders such as thrombosis or thrombophlebitis.
* Fractures, infections and/ or tumor processes.
* Have been treated for plantar fasciitis in the las 4 weeks.
* Previous surgery in the foot
* Pregnancy.
* Communication Disorders.
* Holders of pacemakers or electrostimulators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain scores on the visual analogue scale at 6 weeks in patients with plantar fasciitis. | 6 weeks
  It will evaluate the pain with Visual Analogue Scale in the first step in the first and tenth session. At 6 weeks, a new measurement will be made.

SECONDARY OUTCOMES:
Change in strength scores at 6 weeks from first session in patients with plantar fasciitis. | 6 weeks
  It will evaluate the strength using dynamometer in the first and tenth session. At 6 weeks, a new measurement will be made.
Change in the pain in the Trigger points at 6 weeks from first session in patients with plantar fasciitis. | 6 weeks
  It will evaluate the pain with algometer in the first and tenth session in the plantar muscle. It will measure the change of pain in the Trigger points in the plantar muscle. At 6 weeks, a new measurement will be made .Three measurements will be made and the average data will be recorded.
Change in the functionality of foot and ankle at 6 weeks from first session in patients with plantar fasciitis. | 6 weeks
  It will evaluate the functionality using Foot and Ankle Ability Measure questionnaire (FAAM) in the first and tenth session. At 6 weeks, a new measurement will be made.
Change in the functionality and quality of life of foot and ankle at 6 weeks from first session in patients with plantar fasciitis. | 6 weeks
  It will evaluate the functionality and quality of life using Foot Health Status Questionnaire (FHSQ) in the first and tenth session. At 6 weeks, a new measurement will be made.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Hospital Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Background] Thiagarajah AG. How effective is acupuncture for reducing pain due to plantar fasciitis? Singapore Med J. 2017 Feb;58(2):92-97. doi: 10.11622/smedj.2016143. Epub 2016 Aug 16. PMID 27526703
- [Result] Eftekharsadat B, Babaei-Ghazani A, Zeinolabedinzadeh V. Dry needling in patients with chronic heel pain due to plantar fasciitis: A single-blinded randomized clinical trial. Med J Islam Repub Iran. 2016 Jul 23;30:401. eCollection 2016. PMID 27683642